CLINICAL TRIAL: NCT01341483
Title: Incidence of Male Pudendal Artery Stenosis in Suboptimal Erections Study
Acronym: IMPASSE
Status: Terminated | Type: Observational
Why Stopped: Sufficient information gathered
Sponsor: Medtronic Endovascular (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 00110-229
Record Dates: First submitted 2011-04-20; First posted 2011-04-25 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Erectile Dysfunction Due to Arterial Insufficiency
Keywords: erectile dysfunction; internal pudendal artery; erection; coronary artery disease; peripheral atherosclerotic disease
MeSH Terms: conditions — Erectile Dysfunction; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the proportion of men with known or suspected coronary artery disease (CAD) and/or peripheral arterial disease (PAD) that have angiographic identifiable erectile related artery (ERA) atherosclerotic disease defined as at least one ERA stenosis greater than or equal to 50% (per core lab Quantitative Vascular Analysis - QVA).

DETAILED DESCRIPTION:
Vascular insufficiency is a commonly cited cause of Erectile Dysfunction (ED) and the most common treatments of ED target aspects of the penile vasculature. Initial pharmacotherapy typically focuses on the penile microvasculature; however, surgical revascularization has also been used to treat ED caused by lesions in the internal iliac artery (IIA) and/or internal pudendal artery (IPA) and penile arteries. Anatomically, surgical revascularization connects the inferior epigastric artery to the dorsal artery of the penis or a combination of the dorsal artery and vein of the penis. The pudendal artery or deep artery of the penis is usually not the target of surgical bypass. Recent advances in percutaneous revascularization have sparked interest in penile revascularization to treat ED.

However, as this new percutaneous treatment modality evolves, several important clinical questions remain unanswered. Important among these are what is the normal angiographic anatomy of the erectile related arteries (ERA), and how do angiographic findings correlate with symptoms of ED? Also, how many men could possible benefit from percutaneous revascularization?

The normal IPA anatomy by contrast angiography is not well defined and there are no studies that correlate IPA findings with erectile function. While studies have been done on populations of men with suspected vasculogenic and chronic ED, no study has established the normal angiographic anatomy of the IPA or evaluated the prevalence of angiographic IPA occlusive disease.

Therefore, an angiographic prevalence study will assist in determining the population of men who could potentially benefit from percutaneous treatment of atherosclerotic IPA lesions.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be undergoing coronary or peripheral angiography for suspected or known coronary or peripheral atherosclerotic disease
* Subject must be male ≥ 35 and ≤ 70 years old
* Subject must provide written informed consent before any study-related procedures are performed
* Subject must agree to comply with study procedures and follow-up for the entire length of the study

Exclusion Criteria:

* Subject is unable to safely attempt sexual intercourse secondary to severe cardiac disease or other health condition
* Subject has a life expectancy of < 12 months
* Subject's serum creatinine is > 2.5 mg/dl
* Subject has known aorto-iliac occlusive disease, previous AAA endograft procedure or open surgical procedure
* Subject has history of prostatic carcinoma requiring surgery (i.e., prostatectomy), pelvic radiation, or hormonal/chemotherapy
* Subject has a history of myocardial infarction, stroke, life-threatening arrhythmia, or unstable angina requiring hospitalization within 3 months (90 days) prior to enrollment
* Subject has had exposure to PDE5 inhibitor (per subject's concomitant medication list) within the 72 hours prior to the scheduled baseline angiography
* Subject has a history of renal transplantation
* Subject has a penile implant
* Subject has become unstable or has received a maximum radiation dose, increased procedure time, and/or maximum contrast dose (in the Investigator's opinion) from the primary angiographic procedure that would compromise the safety of the subject by proceeding with enrollment into the IMPASSE study

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of male subjects 35 - 70 years of age undergoing coronary or peripheral angiography and/or intervention for suspected or known coronary or peripheral atherosclerotic disease (CAD or PAD).
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To determine the proportion of men with known or suspected CAD and/or PAD that have angiographic identifiable erectile related artery (ERA) atherosclerotic disease | Baseline through Discharge
  Identifiable ERA disease is defined as at least one ERA stenosis greater than or equal to 50 percent (per core lab Quantitative Vascular Analysis - QVA)

SECONDARY OUTCOMES:
Procedural Safety | 30 Days
  Defined as major adverse event (MAE) rate at 30 days characterized as: 1) Procedure related death (directly related to the ERA DSA portion of the baseline angiography) 2) Occurrence of perineal gangrene or necrosis (penile glans, penile shaft, scrotal or anal) 3) Perineal, penile or anal surgery (including ERA embolization procedures) 4) Renal failure
To determine the proportion of men with atherosclerotic ERA disease who have erectile dysfunction (ED) through 36 months | 36 months
  ED is defined as a urological assessment survey (UAS) of less than or equal to 21
To determine the proportion of men who have atherosclerotic ERA disease and are asymptomatic (i.e., normal erectile function) through 36 months | 36 months
  Normal erectile function is defined as a UAS score greater than 21
To determine the proportion of men who have ED without evidence of atherosclerotic ERA disease through 36 months | 36 months
The predictive capacity of ERA atherosclerosis for potential future cardiovascular events* including ED in men with baseline normal erectile function through 36 months | 36 months
  *Cardiovascular events include - CVA, MI, narrowing of a coronary or peripheral artery resulting in revascularization, new onset hypertension, unstable angina and/or cardiovascular death
The predictive capacity of ED for incident cardiovascular events* compared to men without ED found to have healthy pelvic vasculature (< 50% stenosis in erectile relevant arteries) through 36 months | 36 months
  *Cardiovascular events include - CVA, MI, narrowing of a coronary or peripheral artery resulting in revascularization, new onset hypertension, unstable angina and/or cardiovascular death
Evaluation of the Urological Assessment Survey (UAS) from baseline through the 36 month follow-up period | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Rocha-Singh, MD, Principal Investigator — Prairie Cardiovascular Consultants
Locations (1):
- Prairie Edication and Research Cooperative, Springfield, Illinois, United States